CLINICAL TRIAL: NCT00373373
Title: A Double-blind, Placebo-controlled, Randomized, Multi-center Phase II Trial to Assess the Efficacy of Sorafenib Added to Standard Primary Therapy in Elderly Patients With Newly Diagnosed AML
Brief Title: Efficacy of Sorafenib Added to Standard Primary Therapy in Elderly Patients With Newly Diagnosed AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Bayer (Industry)
Responsible Party: Hubert Serve (Principal Investigator), Klinikum der J.W. Goethe Universität Frankfurt, Med. Klinik II
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KKS/INNERE_A/AML2006; EudraCT Number: 2005-005966-35; Sorafenib in AML
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Sorafenib; Acute Myeloid Leukemia; Flt3; AML; Kinase Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Chemotherapy + Placebo
  Interventions: Drug: Placebo
- B (Active Comparator): Chemotherapy + Sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 2 x 400 mg/d
  Other Names: Nexavar
  Arms: B
Drug: Placebo — Chemotherapy + Placebo
  Arms: A

SUMMARY:
The primary purpose of the study is to determine, whether the addition of Sorafenib to standard chemotherapy in elderly patients with newly diagnosed AML improves treatment results (event free survival).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML (except APL) according to the FAB and WHO classification, including AML evolving from MDS or other hematologic diseases and AML after previous cytotoxic therapy or radiation (secondary AML)
* Bone marrow aspirate or biopsy must contain >= 20% blasts of all nucleated cells, with the exception of AML FAB M6, where >= 30% of non-erythroid cells must be leukemic blasts
* Age >= 61 years
* Informed consent, personally signed and dated to participate in the study
* Male patients enrolled in this trial must use adequate barrier birth control measures during the course of the Sorafenib treatment and for at least 3 months after the last administration of Sorafenib

Exclusion Criteria:

* Central nervous system manifestation of AML
* Cardiac Disease: Heart failure NYHA III° or IV°; active coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Chronically impaired renal function (creatinin clearance < 30 ml/min)
* Chronic pulmonary disease with relevant hypoxia
* Inadequate liver function (ALT and AST >= 2.5 x ULN)
* Total bilirubin >= 1.5 x ULN
* Resting blood pressure (BP) consistently higher than systolic 160 mmHg and/or diastolic 95 mmHg
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardise compliance with the protocol
* Uncontrolled active infection
* Concurrent malignancies other than AML
* Previous treatment of AML except hydroxyurea and up to 2 days <= 100 mg/m²/d cytarabine
* Known HIV and/or hepatitis C infection
* Evidence or history of CNS disease, including primary or metastatic brain tumors, seizure disorders
* Thrombotic or embolic events such as cerebrovascular accident or pulmonary embolism within 1 year of study entry
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* History of organ allograft
* Concomitant treatment with kinase inhibitors, angiogenesis inhibitors and Myelotarg
* Patients with major surgery, open biopsy or significant traumatic injury within 4 weeks of start or first dose
* Serious, non-healing wound, ulcer or bone fracture
* Allergy to study medication or excipients in study medication
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Patients who are not eligible for standard chemotherapy

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Median Event Free Survival of all AML patients

SECONDARY OUTCOMES:
Median Event Free Survival of AML patients with Flt3-ITD mutations
Median Event Free Survival of the patients in each of the four strata (Flt3 Non-ITD/NPM1 WT, Flt3 Non-ITD/NPM1 mut, Flt3 ITD/NPM1 WT, Flt3 ITD/NPM1 mut)
Median Overall Survival of AML patients with Flt3-ITD mutations
Median Overall Survival of all AML patients
Rate of Complete Remission in all AML patients
Rate of Molecular Remission in all AML patients
Toxicity
Evidence of Minimal Residual Disease in all AML patients
Development of Biomarkers indicating the course of disease

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Serve, MD, Principal Investigator — Klinikum der J.W. Goethe Universität Frankfurt, Med. Klinik II
Locations (18):
- Germany (18):
  - Charité Campus Benjamin Franklin, Med. Klinik III, Berlin
  - Klinikum Chemnitz GmbH, Klinik für Innere Medizin III, Chemnitz
  - Klinikum der Universität zu Köln, Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Carl Gustav Carus der TU Dresden, Medizinische Klinik I, Dresden
  - St. Johannes Hospital, Medizinische Klinik II, Duisburg
  - Universitätsklinikum Essen, Zentrum für Innere Medizin, Medizinische Klinik und Poliklinik für Hämatologie, Essen
  - Klinikum der J. W. Goethe-Universität Frankfurt am Main, Medizinische Klinik II, Frankfurt am Main
  - Allgemeines Krankenhaus St. Georg, Hämatologische Abteilung, Hamburg
  - Universitätsklinikum Heidelberg, Med. Klinik V, Heidelberg
  - Klinikum der Johannes Gutenberg Universität, 3. Medizinische Klinik und Poliklinik, Mainz
  - Philipps Universität, Abteilung für Hämatologie, Onkologie und Immunologie, Marburg
  - Klinik für Hämatologie und Onkologie Klinikum Minden, Minden
  - TU München, Medizinische Klinik III, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Münster
  - Klinikum Nürnberg, 5. Medizinische Klinik Einheit für Knochenmarktransplantation, Nuremberg
  - Universität Regensburg, Abteilung für Hämatologie und Internistische Onkologie, Regensburg
  - Robert-Bosch Krankenhaus Stuttgart, Stuttgart
  - Julius-Maximilians-Universität Würzburg, Medizinische Klinik und Poliklinik II, Würzburg